CLINICAL TRIAL: NCT00065273
Title: Severe Aberrant Behavior Among Persons With Mental Retardation. Project III: Behavioral Selectivity of Atypical Neuroleptic Drugs: Effects on Cognitive and Social Behaviors
Brief Title: Atypical Neuroleptic Drugs in People With Mental Retardation/Developmental Delay
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 5P01HD026927 (NIH); 5P01HD026927 (NIH)
Record Dates: First submitted 2003-07-21; First posted 2003-07-22 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-06

CONDITIONS: Mental Retardation; Developmental Delay Disorder
Keywords: Severe aberrant behavior; Risperidone; Clozapine; Haloperidol; Laboratory operant tasks; Simple acquisition procedures; Matching to sample task; Lag sequential analysis
MeSH Terms: conditions — Intellectual Disability; Developmental Disabilities | interventions — Risperidone; Clozapine; Olanzapine

INTERVENTIONS:
Drug: risperidone
Drug: clozapine
Drug: olanzapine

SUMMARY:
Psychiatric drugs are often used to treat behavioral symptoms of mental retardation/developmental delay (MR/DD). These drugs can cause serious side effects. Newer drugs may have decreased side effects. This study will compare new and old drugs used to treat behavioral symptoms in people with MR/DD.

DETAILED DESCRIPTION:
Atypical neuroleptics have fewer extrapyramidal and behavioral side effects than typical neuroleptics. Atypical neuroleptics may also improve social and cognitive functioning. This improvement may be due to reductions in the negative symptoms that are part of the psychosis and psychiatric syndromes or to the improved side effect profile. This study will examine the effects of the atypical neuroleptic drugs risperidone, clozapine, and olanzapine on learning, memory, and social behavior in individuals with MR/DD. A substudy will expand the study to evaluate ecobehavioral measures. The goal of these studies is to assess the behavioral selectivity of atypical neuroleptics by measuring cognitive and social functioning along with targeted aberrant behaviors in individuals under placebo and different doses of drug.

Fifty participants will be randomized to receive risperidone, clozapine, olanzapine, or placebo. Twenty-five of the participants will be drawn from a group receiving typical neuroleptics at the onset of the study. The efficacy of atypical neuroleptics in reducing destructive, aggressive, and stereotypic behaviors in persons with mental retardation will be assessed.

Learning and memory will be measured using laboratory operant tasks. Social and environmental interactions, as well as primary target behaviors, will be directly measured by trained observers. The frequency of specific aberrant behaviors will be determined, along with the conditional probabilities that certain environmental events proceed and follow these behaviors. In the substudy, categories of aberrant behavior will be used to provide information relevant to environmental variables maintaining aberrant behavior; this categorization will improve the determinations of pharmacologic efficacy and will provide a better understanding of the relationship between atypical neuroleptics and environmentally maintained aberrant behavior.

ELIGIBILITY:
Inclusion Criteria

* Primary diagnosis of mental retardation (IQ < 70)
* Scheduled for medication reductions from psychotropic drugs and subsequent placement on risperidone
* Severe self-injury, aggression, property destruction, or stereotypic behavior for 6 months prior to study entry
* No seizures, or seizures under control of medication for previous 2 years

Additional Inclusion Criteria for Substudy

* Participants in the primary study who are available for 2 hour weekly or bi-weekly clinic visits and are able to have observers in their home, school, and/or work environment

Exclusion Criteria

* Degenerative disease that may affect motor or cognitive functioning
* Progressive disease of an organ system
* Advanced age that may produce deteriorating cognitive or motor functioning
* Multiple sensory or motor disabilities that will interfere with seeing the stimuli and responding to the computer

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50
Dates: Start 1998-07; Study Completion 2001-06

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Schroeder, PhD, Principal Investigator — University of Kansas
Locations (1):
- University of Kansas, Lawrence, Kansas, United States

REFERENCES:
- [Background] Valdovinos MG, Napolitano DA, Zarcone JR, Hellings JA, Williams DC, Schroeder SR. Multimodal evaluation of risperidone for destructive behavior: functional analysis, direct observations, rating scales, and psychiatric impressions. Exp Clin Psychopharmacol. 2002 Aug;10(3):268-75. doi: 10.1037//1064-1297.10.3.268. PMID 12233987
- [Background] McAdam DB, Zarcone JR, Hellings J, Napolitano DA, Schroeder SR. Effects of risperidone on aberrant behavior in persons with developmental disabilities: II. Social validity measures. Am J Ment Retard. 2002 Jul;107(4):261-9. doi: 10.1352/0895-8017(2002)1072.0.CO;2. PMID 12069645
- [Background] Zarcone JR, Hellings JA, Crandall K, Reese RM, Marquis J, Fleming K, Shores R, Williams D, Schroeder SR. Effects of risperidone on aberrant behavior of persons with developmental disabilities: I. A double-blind crossover study using multiple measures. Am J Ment Retard. 2001 Nov;106(6):525-38. doi: 10.1352/0895-8017(2001)1062.0.CO;2. PMID 11708938
- [Background] Hellings JA, Zarcone JR, Crandall K, Wallace D, Schroeder SR. Weight gain in a controlled study of risperidone in children, adolescents and adults with mental retardation and autism. J Child Adolesc Psychopharmacol. 2001 Fall;11(3):229-38. doi: 10.1089/10445460152595559. PMID 11642473
- [Background] Hammock R, Levine WR, Schroeder SR. Brief report: effects of clozapine on self-injurious behavior of two risperidone nonresponders with mental retardation. J Autism Dev Disord. 2001 Feb;31(1):109-13. doi: 10.1023/a:1005626100084. PMID 11439749